CLINICAL TRIAL: NCT06405711
Title: To Evaluate the Efficacy and Safety of an Defocus Lens in Slowing the Progression of Myopia：a Prospective Study
Brief Title: To Evaluate the Efficacy and Safety of an Defocus Lens in Slowing the Progression of Myopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY-2023036-2
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Myopia, Progressive
Keywords: myopia; axial length; defocus
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group A (strong higher-order aberrations group) (Experimental): Simultaneous myopic defocus and strong higher-order aberrations lenses
  Interventions: Device: frame lens
- Test group B (medium higher-order aberrations group) (Experimental): Both myopic defocus and medium higher-order aberrations lenses
  Interventions: Device: frame lens
- control groups（HOYA MiYOSMART） (Active Comparator): HOYA MiYOSMART lenses
  Interventions: Device: frame lens

INTERVENTIONS:
Device: frame lens — A randomized block group design was used to randomly assign the included study subjects. The appropriate randomization number and random allocation scheme will be given after enrollment.

SUMMARY:
To confirm the efficacy of DIMS lenses in controlling myopia progression, we planned a prospective, single-centre, randomised, double-blind, controlled, non-inferiority clinical study.

DETAILED DESCRIPTION:
Prior to the trial, subjects signed an informed consent form, screened and qualified subjects were enrolled, and subjects received framed spectacles for correction of myopic refractive error in both eyes, and were fitted with framed spectacles by the investigator according to the standard fitting procedure specified in this protocol. Subjects were randomized to Trial Group A (strong high order aberration group) and Trial Group B (medium high order aberration group) and Control Group (HOYA MiYOSMART).

The index of effectiveness in this clinical trial was to assess the effectiveness of the test group of lenses in slowing the rate of myopia progression by examining the subject's objective optometric values after ciliary muscle paralysis. The basic examination of this clinical trial included slit lamp examination, eye axis examination, fundus examination, corneal topography, best-corrected visual acuity, binocular visual function, refractive status and best-corrected visual acuity after ciliary muscle paralysis, and intraocular pressure measurements, etc. The spectacle fitting was also recorded, as well as the subjective feeling of the subjects when wearing the lenses.

Each subject was followed up for 12 months, and the efficacy and safety of the test product for delaying the progression of myopia was evaluated by the investigator at 1 week ± 1 day (telephone follow-up), 1 month ± 15 days (telephone follow-up), 3 months ± 15 days, 6 months ± 15 days, and 12 months ± 30 days after wearing the lenses.

During the course of this clinical trial, the lenses were replaced due to loss, breakage, change in refraction or poor vision with the lenses, etc., after evaluation by the investigator, and the changes were recorded.

ELIGIBILITY:
Inclusion Criteria:

* The subjects had spherical RE of -1.00 to -6.00 D, astigmatism ≤ 1.50 D, anisometropia ≤ 1.50 D
* the best corrected visual acuity in the left and right eyes subjective optometry is greater than or equal to 1.0

Exclusion Criteria:

* Candidate subjects were excluded from the study if they had strabismus, ocular limitations, or systemic abnormalities affecting vision and ocular motility

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic objective refraction | 12 months
  Cycloplegic objective refraction was measured with an autorefractor (Topcon KR8900, Japan)

SECONDARY OUTCOMES:
Axial Length | 12 months
  Axial length (AL) was measured with an AL-Scan optical biometer (Nidek, Japan)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqin Chen, MD, Principal Investigator — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No